CLINICAL TRIAL: NCT00400166
Title: Recovery Guide Intervention for Recurrent Psychiatric Hospitalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Connecticut State, Department of Mental Health and Addiction Services (Other Government); Eli Lilly and Company (Industry)
Responsible Party: William H. Sledge, M.D.; Director, Yale Psychiatric Hospital; Chair, Yale Department of Psychiatry; George D & Esther S Gross Professor of Psychiatry, Yale University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0607001641
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Last update posted 2009-06-12 (Estimated); Status verified 2009-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Psychotic Depression
Keywords: Peer support; Psychiatric disability; Mutual support; Psychiatric Rehabilitation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Recovery Mentor: peer-based supportive care
  Interventions: Behavioral: Recovery Mentor
- 0 (No Intervention): No Recovery Mentor, services as usual

INTERVENTIONS:
Behavioral: Recovery Mentor — Provided Recovery Mentor services
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether Recovery Guide support services are effective in promoting recovery and social integration among psychiatrically disabled individuals who experience high rates of inpatient hospitalizations.

DETAILED DESCRIPTION:
The paradigm shift in mental health treatment from a deficit-and institution- based framework to a recovery and community integration frame necessitates new models of "case management" practices. The Recovery Guide model is just such a model. Beyond theoretical frameworks, the effectiveness of Recovery Guides has not been well studied. It is the intent of this study to conduct a randomized trial examining the effects of Recovery Guides on community tenure and integration. Furthermore, it is the intent of this study to to establish fidelity criteria.

Comparison(s): Recovery Guide services in addition to treatment as usual, compared to treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Currently admitted in the Yale-New Haven Psychiatric Hospital (YNHPH)
* A history of two or more prior admissions within the past 18 months
* Proficient in the use of the English language
* A DSM-IV diagnosis of Schizophrenia, Schizoaffective Disorder, Psychotic Disorder NOS, or Major Depressive Disorder with Psychotic Features

Exclusion Criteria:

* Inability to give signed, written consent
* Primary DSM-IV diagnosis of substance abuse/dependence

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2006-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Number of hospitalizations | 9 months

SECONDARY OUTCOMES:
Sense of community | Baseline, 3 and 9 months
Motivation for change | Baseline, 3 and 9 months
Social functioning | Baseline, 3 abd 9 months
Hope | Baseline, 3 and 9 months
Self-determination | Baseline, 3 and 9 months
Functional status | Baseline, 3 and 9 months
Treatment relationship | Baseline, 3 and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: William H Sledge, MD, Principal Investigator — Yale University
Locations (1):
- Yale-New Haven Psychiatric Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Derived] O'Connell MJ, Sledge WH, Staeheli M, Sells D, Costa M, Wieland M, Davidson L. Outcomes of a Peer Mentor Intervention for Persons With Recurrent Psychiatric Hospitalization. Psychiatr Serv. 2018 Jul 1;69(7):760-767. doi: 10.1176/appi.ps.201600478. Epub 2018 Apr 16. PMID 29656708
- See also: Yale Program for Recovery and Community Health — http://www.yale.edu/prch